CLINICAL TRIAL: NCT06869915
Title: Prevalence of Neurodevelopmental Disorders in a Homeless Population - Pilot Study
Brief Title: Homelessness and Prevalence of Neurodevelopmental Disorders
Acronym: PRECA'TND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-A01216-41
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Neurodevelopmental Disorders
Keywords: homelessness
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Accommodation, Ocular

STUDY DESIGN:
Intervention Model Description: Every person recruited for the study will undergo a screening phase. If screening is positive, then the person will undergo a diagnostic phase. If screening is negative, the study stops for that person.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Homeless people sheltered in accommodation and social rehabilitation centers (Other): Prevalence (percentage) of ASD, ADHD and IDD in the studied population (homeless people sheltered in accommodation and social rehabilitation centers).
  Interventions: Diagnostic Test: Prevalence (percentage) of ASD, ADHD and IDD in the studied population (homeless people sheltered in accommodation and social rehabilitation centers).

INTERVENTIONS:
Diagnostic Test: Prevalence (percentage) of ASD, ADHD and IDD in the studied population (homeless people sheltered in accommodation and social rehabilitation centers). — This study is an observational prospective multi-centric non interventional study. The focus of the study is a homeless population sheltered in accommodation and social rehabilitation centres. The prevalence of neurodevelopmental disorders in this population will be studied.

SUMMARY:
Introduction & Central question: Psychiatric disorders are highly prevalent in the homeless population, however neurodevelopmental disorders are also at risk of leading to homelessness (Churchard et al., 2018; Casey et al., 2020). Research on this topic is poor in France. This research aims to study the prevalence in France of 3 neurodevelopmental disorders (NDDs) in a homeless population (Autism Spectrum Disorder, Attention Deficit Hyperactivity Disorder and Intellectual Developmental Disorder).

Methods / approach: A 2 phase approach will be used including a screening phase and a diagnosis phase. This research is a pilot study that will include 150 homeless people, over 2 years. The assessment involves combining the results from standardised self-report tools, direct observation and informant-report, thus guaranteeing an objective and thorough diagnosis. This approach gives a better picture of actual behaviour but also a better understanding of the person's development.

OUTCOME: This study will give insight on how to better understand the profile of the homeless population in France, and the prevalence of autism in this population. It will also bring valuable knowledge on how autism and other NDDs can impact one's path in life and lead to homelessness. The results can help develop targeted cares and measures for homeless people with NDDs.

DETAILED DESCRIPTION:
Scientific justification : The main neurodevelopmental disorders (NDDs) are Autism Spectrum Disorder (ASD), Attention-Deficit/Hyperactivity Disorder (ADHD), Intellectual Disability (ID), Specific Learning Disorders and Neurodevelopmental Motor Disorders. This study will focus on three NDDs: ASD, ADHD and ID. Cleaton & Kirby (2018) point out an accumulation and adversity problematic: people with NDDs would accumulate problems over time "in a cascading and cumulative manner" that would lead to adverse medical, psychological and psychosocial outcomes. Many studies have shown the poor outcomes in NDDs. People with ADHD have higher risks of imprisonment (Young & Thome, 2011), poor educational achievement (Fleming et al., 2017), thus unemployment (Halmøy et al., 2009), leading to poor quality of life (Agarwal et al., 2012). ASD has also been linked to unemployment (Bush & Tassé, 2017) or at least to low earnings (Roux et al., 2013), leading to lower quality of life (Ikeda et al., 2014). Unsurprisingly, ID has also been showed to lead to poorer quality of life (Simões & Santos, 2016), because of the higher risk of risky behaviours (Fogden et al., 2016). Thus, all these reasons can lead to social isolation, difficulties in establishing independent living and vulnerability. Homelessness can arise from vulnerability, as much as it can cause it. Homelessness refers to rough sleeping (to sleep in the open air or in places not intended for human habitation, Crisis, 2017.), but also to people who sleep in adapted sleeping places but who do not have any official title to the accommodation (Fazel et al., 2014). A recent French study (Laporte et al., 2018) concluded that more than 30% of homeless people suffer from mental health disorder (13.2% would have psychosis, 12.3% severe anxiety disorder, 6.7% severe mood disorder). There is an increasing number of studies linking mental health and homelessness, however research on NDDs and homelessness is still rather poor. Two British studies have found a high prevalence of ASD among homeless adults. They explain this prevalence by the difficulty for these people to get and keep a job (Churchard et al., 2018; Kargas et al., 2019). Kargas et al., 2019 have found that 18.5% of their homeless population presented with scores superior to 7 at the AQ-10, consistent with high levels of autistic traits. A prospective study has shown that out of 135 children with ADHD, 23.9% have known homelessness at least once in their adult life (García Murillo et al., 2016). Riglin et al., (2023) explain that 20% of young socially precarious adults would suffer from ADHD. Durbin et al., (2018) claim that the prevalence of ID in a homeless population would be between 12 and 39%, this is corroborated by Brown & McCann., (2021) who point out that 10 to 39% of homeless people would have an ID. These international studies point out the probable links between homelessness and NDDs, however this field of research is lacking in France.

Main aim of the study : to study the prevalence of the following 3 NDDs (ASD, ADHD, IDD) in a homeless population received in accommodation and social rehabilitation centres

Secondary aims :

1. To compare the social, demographic, medical and judicial characteristics of homeless people with NDD and homeless people without NDD.
2. To research the frequency of traumatic brain injury, coma and epilepsy in this homeless NDD population.

Methodology :

This study is an observational prospective multi-centric non interventional study.

1. Pre-inclusion: a neuropsychologist will give all the information concerning the study to the patients.
2. Screening :

   * 1st Visit (V1) (1h30) : carried out by a neuropsychologist : written and signed consent for the study and thorough screening for NDDs
   * 2nd visit (V2) (1h30) : carried out by a psychiatrist only after a positive screening for one or more NDDs. The psychiatrist will then carry out a developmental anamnesis and then carry out the necessary diagnostic tools.
   * Visit with a social worker (45 min): carried out by the psychiatrist or the neuropsychologist in order to collect more specific information on the daily life of the person and help in the diagnostic process.
3. End of the research and diagnostic announcement (V3): (45 min), carried out by the psychiatrist, with the participants who did V1 and V2. The psychiatrist will give the results and the diagnosis if pertinent. Specific care and health issues will be discussed.

Population studied: Homeless people sheltered in accommodation and social rehabilitation centres

ELIGIBILITY:
Inclusion Criteria:

* Homeless people sheltered in accommodation and social rehabilitation centers
* Over 18 years of age
* Who speak French
* who have given then written informed consent

Exclusion Criteria:

- Every person who hasn't given their written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence (percentage) of ASD, ADHD and IDD in the studied population (homeless people sheltered in accommodation and social rehabilitation centers). | 4 months
  For each NDD here are the scores and tools used :
  ASD :
  * AQ-10 cut-off score
  * CAT-Q cut-off score(Camouflage of Autistic Traits Questionnaire)
  * Glasgow questionnaire : standard score deviations
  * DATHi (DSM-5 Autistic Traits in the Homeless Interview) : cut-off score
  ADHD:
  * ADHD Self-report (ASRS) : cut-off score
  * Diagnostic Interview for Adult ADHD (DUVA-5): cut-off score
  * ASRS - Observer : cut-off score
  IDD:
  * Raven matrices: score
  * Vineland Adaptive Behaviour Scale (2nd edition): cut-off score

SECONDARY OUTCOMES:
Demographic information | 4 months
  Age, education, professional career, time without a home and duration of homelessness The measures will be in number of weeks, months or years
Judicial information | 4 months
  Record of conviction, sentences and imprisonment
Medical Record | 4 months
  Medical treatments, care, mental health issues
Drug abuse | 4 months
  History of drug abuse, which drugs, quantities
History of traumatic brain injury, epilepsy and coma | 4 months
  History of traumatic brain injury (yes / no); coma (yes /no); epilepsy (yes / no)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline DEMILY, MdPh, Principal Investigator — VINATIER HOSPITAL
Locations (1):
- Hopital Vinatier, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No